CLINICAL TRIAL: NCT05199896
Title: Touching the World With a (Blind) Cane: Cognitive and Neural Processes
Brief Title: Touching the World With a Cane: Cognitive and Neural Processes
Acronym: TOOL_TOUCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL21_0882
Record Dates: First submitted 2022-01-04; First posted 2022-01-20 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Visual Impairment; Healthy
Keywords: Blind/Non-sighted; Healthy subject; fMRI; EEG
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- All protocols (behavioral and EEG and fMRI) (Experimental): If participants accepts (non-sighted participants and Healthy volunteers), they will carry out the behavioral protocol and the EEG protocol and fMRI protocol.
  Interventions: Behavioral: Behavioral protocol; Device: EEG protocol; Device: fMRI protocol
- Behavioral protocol and EEG protocol (Experimental): Participants who agree to participate in only one of the experiments (EEG or MRI) will be randomly (by a randomization list) assigned to either the EEG or fMRI type of study in each subgroup.
  All participants (non-sighted participants and Healthy volunteers) will do the behavioral session and at least one EEG or MRI session depending on randomization.
  Interventions: Behavioral: Behavioral protocol; Device: EEG protocol
- Behavioral protocol and fMRI protocol (Experimental): Participants who agree to participate in only one of the experiments (EEG or MRI) will be randomly (by a randomization list) assigned to either the EEG or fMRI type of study in each subgroup.
  All participants (non-sighted participants and Healthy volunteers) will do the behavioral session and at least one EEG or MRI session depending on randomization.
  Interventions: Behavioral: Behavioral protocol; Device: fMRI protocol

INTERVENTIONS:
Behavioral: Behavioral protocol — A touch sensitive computer screen either displaying a downscaled (45cm long) image of the rod (for the sighted), or supporting a same sized wooden rod (for the blind), will be placed on the table in front of the participant to record their localization performance. They will be instructed to use their left index fingertip to indicate on the image of the screen (for sighted) or on the wooden rod (for the blind) the position where they have felt the touch provided to the 90 cm long they held in their right dominant hand. Participants will wear a headset playing white noise to prevent any auditory localization cues when the long rod will be touched. The rod will be touched by a computer controlled solenoid. Thus, participants will respond with a hand gesture on the image or rod and will be asked to validate the position by pressing a foot-pedal with their left foot.
Device: EEG protocol — The EEG protocol will be similar as the behavioral one described above, with the distinction of taking place in two separate sessions: one where the rod are touched, and one where their hand is touched. The participant will hold a rod in each hand and he will have to indicate on which rod he felt the touch.
  Additionally electrophysiological responses will be continuously recorded using a 65 channel ActiCap system (Brain Products).
  Arms: All protocols (behavioral and EEG and fMRI); Behavioral protocol and EEG protocol
Device: fMRI protocol — The same behavioral task and procedures of the behavioral protocol described above will be applied, adapted to take into account the constraints posed by the magnetic environment of the MR scanner. The participant will be placed on the scanner bed and provided with earphones that will both protect against the noise of the machine (80dB) and ensure a continuous communication with the participant.
  During the fMRI sessions, the participant will solve the same rod localization behavioral task while we will record brain activations by measuring the brain oxygen level dependent signal via Echo Planar Imaging sequences. We will use an MRI compatible tactile stimulator to touch the hand-held rod and participants location judgement will be recorded by using an MRI-compatible tablet, positioned on their abdomen, where the participant will have to indicate the judged position.
  Arms: All protocols (behavioral and EEG and fMRI); Behavioral protocol and fMRI protocol

SUMMARY:
The use of tools is ubiquitous in our lives and allows us to expand the sensorimotor capacities of our body. Much research has been done on the subject in sighted people over the past decades. This work has mainly focused on the motor aspect of using the tool, neglecting the sensory aspect. However, any action involving a tool carries sensory information, for example in the use of the white cane by blind people. 26% (> 200,000) of blind people in France use a white cane to get around. By sweeping the cane on the ground, they use it as a sensorimotor extension of their body to extract information from the environment in order to locate a pedestrian crossing or possible obstacles. While it is well established that the tools increase the user's motor skills, we have only just begun to clarify how they also function as sensory extensions of the user's body and how this phenomenon is potentially dependent on constant use of the tool to compensate for a missing sense, as is the case with blind people using a cane. The aim of this study is to fill this important gap in our knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, aged 18 to 60 years old
* Give an informed consent by signature
* Be part of the national health security system (registered to the Securité Sociale)
* do not confuse his right and his left

Specific of the non-sighted participants:

* Loss of vision happened at birth or 3-to 5 years later in life
* Must have a visual acuity inferior or equal to 4/10
* Be with a close relation for read information letter and sign the consent form if needed

Exclusion Criteria:

* A person presenting an history of neurological, psychiatric or linguistic problems cannot be admitted
* Assumption of psychotropic drugs
* Pregnancy or breast-feeding woman
* A person under legal tutoring
* A person under care in other medical structure for reasons different from those of this research
* A person under administrative or judiciary contention
* A person who is not eligible to a MRI-exam according to the following criteria cannot be admitted to the experiments including MR acquisitions :

  * Have a neurological, cardiac (battery) or defibrillator pacemaker
  * Have a cardiac prosthesis (valve, stent...) or vascular prosthesis
  * Have intracranial clips or clamps
  * Carry a bypass of the cerebrospinal fluid
  * Having metallic splinters in the eyes
  * Wear metal prostheses (teeth, knees)
  * Wear an infusion pump or system
  * Be claustrophobic or have respiratory problems
  * Have metal tattoos close to the head
  * Have permanent make-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Perceived location | 90 minutes
  Tactile stimulus will be applied on a tool (a rod). Subject should determine the exact spatial location of the stimulus.
  This will be measure at each stimulation.

SECONDARY OUTCOMES:
Brain activity | 6 hours
  Brain oscillatory activity and the somatosensory evoked potentials during the realization of experimental tasks on EEG.
  Two sessions of about 3 hours are necessary for the EEG acquisition.
Brain activity | 3 hours
  Measuring the brain oxygen level dependent (BOLD) signal during the realization of experimental tasks on fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Equipe IMPACT du CRNL, Bâtiment INSERM, Bron, France

IPD SHARING:
Plan to Share IPD: No